CLINICAL TRIAL: NCT07033806
Title: TABATA EXERCISE IMPROVED NON-DOMINANT LOWER EXTREMITY STRENGTH IN NORDIC SKIERS
Acronym: BOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Doç.Dr. Emrah AYKORA, Assoc. Prof., Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: TYL-2022-3923; TYL-2022-3923 (Other Grant/Funding Number: Çanakkale Onsekiz Mart University Experimental Research Coordination Unit)
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Laterality; Exercise
Keywords: Nordics, ski runners, laterality, non-dominant extremity, Tabata exercise, training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: tabata exercise and normal exercise
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Tabata protocol
  Interventions: Other: Exercise Tabata Protocol
- Exercise (Experimental): Tabata protocol
  Interventions: Other: Exercise Tabata Protocol

INTERVENTIONS:
Other: Exercise Tabata Protocol — more effective

SUMMARY:
Background: Laterality in athletes presents the preference to overuse extremities, which weakens the non-used parts, resulting in an uneven power distribution and body imbalance. There is a lack of knowledge and studies to elucidate those drawbacks. Qualitative and high-intensity exercise for the non-dominant extremity has the potential to avoid laterality and enhance the whole-body performance for the race.

ELIGIBILITY:
Inclusion Criteria:

* having no existing disability or severe injury during the last 5 years, having no existing psychological disorders.

Exclusion Criteria:

* having existing disability or severe injury during the last 5 years, having existing psychological disorders.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Number of Steps and Cross-Continuity | 3 months
  Single leg skating steps numbers were measured

SECONDARY OUTCOMES:
muscle strength | First 3 months
  The muscle strength was evaluated from three major muscles in every exercise session

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided